CLINICAL TRIAL: NCT02534740
Title: A Phase 1, Open-Label, Randomized, Single Dose Study To Estimate The Relative Bioavailability And Food Effect Of PF-06291826 (Tafamidis) Following Administration Of New Soft Gelatin Capsule Oral Formulations In Healthy Subjects
Brief Title: A Study Comparing Amounts of Tafamidis In The Blood With Or Without Food
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: B3461052; 2015-002315-15 (EudraCT Number)
Record Dates: First submitted 2015-08-25; First posted 2015-08-28 (Estimated); Last update posted 2015-12-22 (Estimated); Status verified 2015-12

CONDITIONS: Healthy
MeSH Terms: interventions — tafamidis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- 4 soft gel capsules of 20 mg tafamidis meglumine (Experimental)
  Interventions: Drug: tafamidis
- 48.8 mg tafamidis soft gel capsule formulation 1 (Experimental)
  Interventions: Drug: tafamidis
- 48.8 mg tafamidis soft get capsule formulation 2 (Experimental)
  Interventions: Drug: tafamidis
- 61 mg tafamidis soft gel capsule formulation 1 (Experimental)
  Interventions: Drug: tafamidis
- 61 mg tafamidis soft gel capsule formulation 2 (Experimental)
  Interventions: Drug: tafamidis

INTERVENTIONS:
Drug: tafamidis — relative bioavailability
  Arms: 4 soft gel capsules of 20 mg tafamidis meglumine; 48.8 mg tafamidis soft gel capsule formulation 1; 48.8 mg tafamidis soft get capsule formulation 2
Drug: tafamidis — fasted
  Arms: 61 mg tafamidis soft gel capsule formulation 1; 61 mg tafamidis soft gel capsule formulation 2
Drug: tafamidis — fed
  Arms: 48.8 mg tafamidis soft gel capsule formulation 1; 48.8 mg tafamidis soft get capsule formulation 2

SUMMARY:
This is a 2 part study. In part 1 of the study, 3 different formulations of the same dose of tafamidis will be compared. Subjects will be fasted for each test and every subject will test all 3 different formulations. After swallowing tafamidis, tafamidis blood concentrations will be measured periodically for 6 days. After 14 days, subjects will take a different formulation of tafamidis and tafamidis blood concentrations will be measured periodically for 6 days. After another 14 days, the last formulation will be tested in the same way. In part 2 of the study, depending on the results of part 1, either none, one or 2 of the formulations tested in part 1 will be tested comparing the same formulation when given either with or without food. Additionally, depending on the results of part 1 of the study, different doses of the formulations may be compared.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males or females of non-child bearing potential.
* Body Mass Index (BMI) of 17.5 to 30.5 and total body weight more than 50 kg (110 lbs).

Exclusion Criteria:

* Blood pressure at screening visit of greater than 140 mm Hg (systolic) or 90 mg Hg (diastolic).
* Use of prescription or nonprescription drugs supplements within 7 days prior to 7 days of the study.
* Pregnant female subjects; breastfeeding female subjects; male subjects with partners currently pregnant; male subjects able to father children who are unwilling or unable to use a highly effective method of contraception.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2015-09; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Area under the concentration-time Curve (AUC) | 120 hours
Maximum Observed Plasma Concentration (Cmax) | 120 hours

SECONDARY OUTCOMES:
Area Under the Curve From Time Zero to Last Quantifiable Concentration (AUClast) | 120 hours
Time to Reach Maximum Observed Plasma Concentration (Tmax) | 120 hours
Plasma Decay Half-Life (t1/2) | 120 hours
Area Under the Curve from Time zero to infinity | 120 hours

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Clinical Research Unit, Brussels, Belgium